CLINICAL TRIAL: NCT05147116
Title: The Effects of Repeated Moderate Overnight Normobaric Hypoxia on Glucose Homeostasis, Appetite, Body Weight, Inflammation and Oxidative Stress in Individuals With Type 2 Diabetes Mellitus
Brief Title: The Effect of Hypoxia on Type 2 Diabetes and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Bournemouth University (Other); University College, London (Other); University of Cambridge (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Ant Shepherd, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 009AS
Record Dates: First submitted 2021-11-08; First posted 2021-12-07 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Sleep

STUDY DESIGN:
Intervention Model Description: Single blind, randomized, balanced, crossover design study
Who Masked: Participant
Masking Description: Participants will undergo both the hypoxia and sham conditions and will be blinded to the conditions in which they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxia 15% O2 (Experimental): Participants will sleep in a tent for 10 nights in hypoxia.
  Interventions: Other: Sleeping in a tent
- Sham (room air) 21% 02 (Sham Comparator): Participants will sleep in a tent for 10 nights in normoxia.
  Interventions: Other: Sleeping in a tent

INTERVENTIONS:
Other: Sleeping in a tent — Participants will spend 10 consecutive nights of sleeping in a tent

SUMMARY:
The number of people with type 2 diabetes mellitus (T2DM) continuing to rise, this pandemic is expected to reach 700 million people by 2045. T2DM is a metabolic condition characterized by progressive insulin resistance and chronic hyperglycemia (high blood glucose concentrations). Hyperglycaemia increases the risk of both micro- and macrovascular damage, whilst interventions that reduce blood glucose mitigate this risk. Weight loss, achieved through exercise and dietary modification, is effective at reducing hyperglycaemia. However, despite the clear benefits of exercise and weight loss, diverse psychological, sociological and logistical factors can make it difficult for some individuals with T2DM to initiate, or adhere to, these lifestyle interventions. Alternative approaches to treatment are therefore required.

The purpose of this research project is to investigate whether 10-days of overnight exposure to moderate hypoxia is effective at improving blood glucose control in individuals with T2DM and to provide insight into the physiological mechanisms responsible for any beneficial effects.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a metabolic condition characterized by progressive insulin resistance and chronic hyperglycemia (high blood glucose concentrations). Hyperglycaemia increases the risk of both micro- and macrovascular damage, whilst interventions that reduce blood glucose mitigate this risk. Weight loss, achieved through exercise and dietary modification, is effective at reducing hyperglycaemia. However, despite the clear benefits of exercise and weight loss, diverse psychological, sociological and logistical factors can make it difficult for some individuals with T2DM to initiate, or adhere to, these lifestyle interventions. With the number of people with T2DM continuing to rise, this pandemic is expected to reach 700 million people by 2045. Thus, there is a clear need for cost-effective interventions that can effectively improve glycaemic control in people with T2DM and which people will adhere to.

A simple exposure to a lowered concentration of inspired oxygen (i.e. hypoxia) may represent such an intervention. In addition to the beneficial effects on glucose homeostasis that have been reported following a single acute hypoxic exposure, repeated intermittent, or continuous, hypoxic exposure may also have therapeutic potential in individuals with T2DM. In rodent models, daily hypoxic exposures returned fasting blood [glucose] to normal levels and increased glucose transporter 4 translocation in mice with T2DM. Similar effects on glucose homeostasis have been shown in overweight humans and those with insulin resistance, (during intermittent hypoxic training) which was explained, at least in part, by reduction in body mass (~ 1.2 kg).

The mechanisms underpinning the improved glycaemic control in response to hypoxia are likely multifactorial. Specifically, our objective is to assess a novel therapeutic intervention for the treatment and management of T2DM which overcomes many of the barriers to uptake and adherence that are associated with some lifestyle interventions such as exercise and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Males and post-menopausal women with T2DM (as diagnosed with the WHO criteria).

Exclusion Criteria:

* Individuals with contraindications to hypoxic exposure (e.g. obstructive sleep apnoea, extant cardiac conditions or on medications such as SGLT2 inhibitors or PPAR antagonists).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Shepherd, PhD, Principal Investigator — University of Portsmouth
Locations (1):
- Anthony Shepherd, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The individual data set that is used for statistical analysis will be uploaded to our university repository and a DOI added to the paper upon publication.
Time Frame: Upon publication - no plan to remove.
Access Criteria: Dataset is open access from the URL below.
URL: https://researchportal.port.ac.uk/en/datasets/hypoxiat2dmdata

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypoxia 15% O2 - Sham (Room Air) 21% O2: Participants will sleep in a tent for 10 nights in hypoxia. They will then have a 3 month washout, crossover and do another 10 nights but in normoxia.
- Sham (Room Air) 21% 02 - Hypoxia 15% O2: Participants will sleep in a tent for 10 nights in normoxia. They will then have a 3 month washout, crossover and do another 10 nights but in hypoxia.
Period: Overall Study
Arm/Group | Hypoxia 15% O2 - Sham (Room Air) 21% O2 | Sham (Room Air) 21% 02 - Hypoxia 15% O2
Started | 8 | 6
Completed | 8 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: As this is a within-subject, repeated measures RCT, participant characteristics are presented as one.
Arm/Group | Total
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 13
Height [Mean (Standard Deviation); unit: m] | 1.72 (0.09)
Mass [Mean (Standard Deviation); unit: kg] | 87.5 (14.6)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.7 (3.9)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 61.1 (14.1)
T2DM duration [Mean (Standard Deviation); unit: years] | 9.3 (7)
SBP [Mean (Standard Deviation); unit: mmHg] | 132 (13)
DBP [Mean (Standard Deviation); unit: mmHg] | 80 (11)

OUTCOME MEASURES:

1. Primary Outcome: Δ Mean AUC (Area Under the Curve) Plasma [Glucose]
Description: Does 10 days of overnight hypoxia change AUC during a oral glucose tolerance test. Units for AUC are AU (arbitrary units) which have been derived from the trapezoidal method and have been published as such. Trapezoidal method: AUC = Δx ((y0/2)+y1+y2+y3+...+(yn/2)).
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: Assessed on all outcome visits (2,3,4&5) across an 8 week period. Δ from pre-post hypoxia visits are calculated and compared to Δ from pre-post sham visits.
Measure: Mean (Standard Deviation); unit: mmol.min.L-1
Groups:
- Sham (Room Air) 21% O2: Participants will sleep in a tent for 10 nights in normoxia.
  Sleeping in a tent: Participants will spend 10 consecutive nights of sleeping in a tent
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 11 | 11
mmol.min.L-1 | -17.7 (237.7) | 54.9 (226.1)

2. Secondary Outcome: Δ Body Mass
Description: Does 10 days of overnight hypoxia change body mass - assessed via DXA.
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: as for outcome 1
Population: Within-subject cross-over trial. Total still did not exceed 13.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Hypoxia 15% O2: Participants will sleep in a tent for 10 nights in hypoxia. They will then have a 3 month washout, crossover and do another 10 nights but in normoxia.
- Sham (Room Air) 21% O2: Participants will sleep in a tent for 10 nights in normoxia. They will then have a 3 month washout, crossover and do another 10 nights but in hypoxia.
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 13 | 12
kg | 0 (0.9) | -0.7 (1)

3. Secondary Outcome: Δ Total Minutes of Physical Activity (Light, Moderate, Moderate to Vigorous Physical Activity).
Description: Does 10 days of overnight hypoxia change physical activity - assessed via wrist worn accelerometry.
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: as for outcome 1
Population: Within-subject crossover trial. Therefore total is still 10.
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 10 | 10
min | 170 [103 to 237] | 183 [116 to 250]

4. Secondary Outcome: Δ Sleep Efficiency (Percentage of Time Spent Asleep While in Bed)
Description: Does 10 days of overnight hypoxia change sleep - assessed via wrist worn accelerometry.
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: as for outcome 1
Population: Within-subject crossover trial. Therefore total is still 10.
Measure: Median (Inter-Quartile Range); unit: % of time spent asleep while
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 10 | 10
% of time spent asleep while | 88 [79 to 97] | 86 [78 to 94]

5. Secondary Outcome: Δ IL-6
Description: Does 10 days of overnight hypoxia change IL-6.
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: as for outcome 1
Population: Within-subject crossover trial. Therefore total is still 12.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 12 | 12
pg/mL | 1.06 [-1.66 to 3.78] | -0.55 [-2.08 to 0.98]

6. Secondary Outcome: Δ TNFɑ
Description: Does 10 days of overnight hypoxia change TNFɑ.
  Due to the study design being a randomised crossover control trial, the results for visits 2 and 3, and, 4 and 5, have been unrandomized into the delta of pre-post hypoxia and sham interventions. Visits 2 and 4 represent baseline compared to visit 3 and 5 respectively.
Time Frame: as for outcome 1
Population: Within-subject crossover trial. Therefore total is still 12.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
Number analyzed (Participants) | 12 | 12
pg/mL | 0.66 [-2.06 to 3.38] | 0.61 [-1.75 to 2.97]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Within-subject crossover trial. Therefore total is still 22 (i.e. the number of individuals who took part in at least visit 1.)
Groups:
- Sham (Room Air) 21% O2: Participants will sleep in a tent for 10 nights in normoxia.
Arm/Group | Hypoxia 15% O2 | Sham (Room Air) 21% O2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT05147116/Prot_SAP_000.pdf